CLINICAL TRIAL: NCT00035048
Title: A Double-Blind, Placebo-Controlled, Multicenter Study of the Long-Term Efficacy of MK0869 in the Maintenance of Antidepressant Effect in Geriatric Outpatients With Major Depressive Disorder
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-068)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-068; Formally-3N25; MK0869-068; 2006_406
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: aprepitant
  Other Names: MK0869
Drug: Comparator: placebo (unspecified)

SUMMARY:
A clinical study to determine the efficacy and safety of an investigational medication (MK0869) in the treatment of depression.

DETAILED DESCRIPTION:
The duration of treatment is 10 weeks.

ELIGIBILITY:
Patients with Major Depressive Disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 540 (Actual)
Dates: Start 2001-11-21 (Actual); Primary Completion 2003-12-29 (Actual); Study Completion 2003-12-31 (Actual)

PRIMARY OUTCOMES:
HAMD-17 score </= 10 after 10 weeks; maintenance of antidepressant effect for 6-10 months; tolerability | After 10 weeks & 6-10 months

SECONDARY OUTCOMES:
CGI-S score change from Week 10 at Month 6; HAMD-17 total score change from Week 10 at Month 6; MADRS total score change at Month 6, HAMA total score change at Month 6 | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html